CLINICAL TRIAL: NCT04425161
Title: Role of "Central Venous-to-Arterial Carbon Dioxide" to "Arterial-to-Central Venous Oxygen Content" Ratio, as a Marker of Anaerobic Metabolism in Septic Shock
Brief Title: Ratio of ''Central Venous-to-Arterial Co2 Gap'' to ''Arterial-to-Central Venous O2 Content Gap'' in Septic Shock
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ahmed Atta Ahmed Elsawy, Principal Investigator, Ain Shams University
Other Study IDs: FMASU MD 1322018
Record Dates: First submitted 2020-06-06; First posted 2020-06-11 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Septic Shock
Keywords: sepsis; PCO2 gap; PCO2 gap/ O2 content gap
MeSH Terms: conditions — Shock, Septic; Sepsis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- VO2 ≥15 %: This group is classified based on increased oxygen consumption (VO2) ≥15 % by volume expansion in fluid responders
  Interventions: Other: Fluid challenge (0.9 % NaCl)
- VO2 <15 %: This group is classified based on increased oxygen consumption (VO2) < 15 % by volume expansion in fluid responders
  Interventions: Other: Fluid challenge (0.9 % NaCl)

INTERVENTIONS:
Other: Fluid challenge (0.9 % NaCl) — 500 ml Fluid challenge of (0.9 % NaCl) will be given

SUMMARY:
The high ratio of "central venous to arterial carbon dioxide" to "arterial to central venous oxygen content " is associated with elevated lactate in patients with septic shock.

So, the aim of the present study is to evaluate the ratio of "central venous-to-arterial CO2 tension or content" to "arterial-to-venous O2 content'' as an indicator of anaerobic metabolism in septic shock.

DETAILED DESCRIPTION:
This is a prospective single center observational study that will be conducted in adult intensive care unit of Ain Shams University After being approved by local institutional ethic committee (Ain Shams University, Egypt). Informed consent was obtained from each participant's next of kin. The investigator will study mechanically ventilated participants. the attending physician's decision is to give IV fluids to participants due to the presence of at least one clinical sign of inadequate tissue perfusion due to septic shock : (a) systolic arterial pressure <90 mmHg, mean arterial pressure <65 mmHg, or the need for vasopressor infusion; (b) skin mottling; (c) lactate level >2 mmo/L; or (d) urinary output <0.5 mL/kg/h for ≥2 h. Jugular central venous and arterial catheters will be in place by the attending physician. Investigator will confirm the position of the tip of the central venous catheter in the superior vena cava or upper part of the right atrium on chest radiograph. Participants will be monitored by Flo Trac device as a part of routine management in local ICU.

A first set of measurements will be performed, including hemodynamic and tissue oxygenation variables (heart rate, mean arterial pressure, cardiac index (CI), oxygen delivery (DO2), oxygen consumption (VO2), Central venous oxygen saturation (ScvO2), arterial lactic acid level, central venous to arterial carbon dioxide tension difference (∆PCO2), central venous to arterial CO2 content difference (∆ContCO2), arterial-to-central venous oxygen content difference (∆ContO2), ∆ContCO2/∆ContO2 ratio and ∆PCO2/∆ContO2 ratio. 500 ml of isotonic saline 0.9% will be infused to the participants via a specific venous line over 15 minutes. Immediately after volume expansion, a second set of the previous measurements will be recorded. Ventilation parameters, Norepinephrine dose and sedation drugs will be kept constant during the fluid challenge.

After fluid challenge, Participants with an increase in cardiac index ≥15% will be defined as fluid responders. Fluid responders will be divided into 2 groups based on increase in oxygen consumption (VO2) ( < or ≥15%).

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years.
2. Suspected infection focus
3. Mean blood pressure <65 mmHg, or required vasopressor infusion.
4. Lactic acid level >2 mmol/l.
5. Mechanically ventilated patients.

Exclusion Criteria:

1. Age equal or less than 18 years.
2. Pregnant women.
3. Liver cirrhosis Child-Pugh C.
4. Chronic obstructive pulmonary disease.
5. Previous episode of septic shock within the last 3 months.
6. Patients with a contraindication to volume expansion.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients who will be admitted to intensive care units and eligible for the study.
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the change of the ratio of "central venous-to-arterial CO2 tension or content" to "arterial-to-central venous O2 content" as an effective marker to indicate anaerobic metabolism in septic shock. | Measurements will be taken immediately before and immediately after volume expansion
  To evaluate the change of the ratio of "central venous-to-arterial CO2 tension or content" to "arterial-to-central venous O2 content" between immediately before and Immedialey after volume expansion to indicate anaerobic metabolism in septic shock.

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed A Elsawy, Master, Principal Investigator — Ain Shams University; Ayman M Kamaly, Professor, Study Director — Ain Shams University
Locations (1):
- AinShams, Cairo, Egypt